CLINICAL TRIAL: NCT03075007
Title: White Matter Hyperintensities in Aging and Dementia
Brief Title: Brain Vascular Disease in Aging and Dementia
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Adam Brickman, Associate Professor of Neuropsychology, Columbia University
Other Study IDs: AAAR1423; 2R56AG034189-06A1 (NIH)
Record Dates: First submitted 2017-03-06; First posted 2017-03-09 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Alzheimer Disease; White Matter Hyperintensities; Dementia; Aging
Keywords: Alzheimer Disease; Aging; Dementia; PET
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — 4-(N-methylamino)-4'-(2-(2-(2-fluoroethoxy)ethoxy)ethoxy)stilbene; Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group A: All participants will undergo an amyloid PET scan with Florbetaben F 18 contrast as well as a transcranial Doppler ultrasound.
  Interventions: Radiation: Florbetaben F18; Procedure: Transcranial Doppler

INTERVENTIONS:
Radiation: Florbetaben F18 — 10Meq of Florbetaben F 18 via intravenous injection is to be used. Visit duration is approximately 3 hours.
Procedure: Transcranial Doppler — All participants will undergo Doppler ultrasonography that measures the velocity of blood flow through the brain's blood vessels. Visit duration is approximately 45 minutes and will be scheduled for either the same day or another day as the PET scan.

SUMMARY:
This study examines the factors that may drive the relationship between vascular disease and Alzheimer's Disease (AD) in a large, longitudinal, multi-ethnic community-based cohort study of older adults in northern Manhattan, New York. In past research, the investigators demonstrated that accumulation of brain vascular disease is associated with risk for development of AD. The study now extends the research to examine how brain vascular disease and AD interact. In this pilot study, the investigators will obtain positron emission tomography (PET) scans to measure amyloid (one of the protein pathological markers of AD) from participants in an ongoing community-based study of aging and dementia (WHICAP). The study will include subjects who are already enrolled in the parent project. Further, this study will enroll both subjects who have never been evaluated with PET scans and those who received a previous baseline PET scan. The study plans to obtain approximately 30 repeat amyloid PET scans and 20 baseline PET scans. The investigators will also conduct transcranial Doppler studies to measure blood flow in the participants with amyloid PET scans. The potential benefits to society should be considerable if this study reveals new information about risk factors for or contributions to AD.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is one of the most devastating international public health epidemics. There are currently no effective disease-modifying or preventative strategies. Current pathogenic models emphasize a single pathway of disease pathogenesis, but underestimate the contribution of small vessel cerebrovascular disease, which manifests primarily as white matter hyperintensities (WMH) on T2-weighted magnetic resonance imaging (MRI). Understanding of the factors that drive the relationship between vascular disease and AD remains elusive; vascular factors may be independent sources of dysfunction that contribute additively to clinical expression, they may interact mechanistically with AD pathology, and/or they may relate to each other because of a shared association with a third set of factors. These issues are particularly relevant among ethnic/racial minorities, who are at much greater risk for clinical AD, have more severe cerebrovascular disease, but appear to have similar levels of AD pathology compared with Whites.

The proposed research examines these factors in a large, longitudinal, multi-ethnic community-based cohort study of older adults in northern Manhattan, New York. The investigators demonstrated that accumulation of WMH, particularly in parietal lobes, predicts incident AD, and is associated with the presence of cerebral microbleeds, an indicator of cerebral amyloid angiopathy. The investigators extend the research to examine mechanistic interactions between cerebrovascular disease and AD. The preliminary data suggest that individuals with evidence of fibrillar amyloidosis have increased parietal lobe WMH and that hemodynamic markers of autoregulatory dysfunction are associated with both WMH and amyloid deposition, which in turn interact to promote the clinical expression of AD. These findings are buffered by new data that establish WMH as a core feature in autosomal dominant forms of AD. In this pilot study, the investigators propose to obtain cross-sectional and longitudinal MRI and amyloid PET data from participants in WHICAP.

ELIGIBILITY:
Inclusion Criteria:

* current participant in WHICAP (Washington Heights/Inwood Columbia Aging Project)
* subject previously participated in baseline MRI sub-study
* post-menopausal

Exclusion Criteria:

* allergic to Florbetaben
* claustrophobic
* liver problems
* history of epilepsy/seizures
* pre-menopausal
* serious medical conditions

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential participants are recruited from a list of active members in the Washington Heights/Hamilton Heights/ Inwood Columbia Aging Project, known as WHICAP (CU IRB# AAAO9804), who previously completed a repeat MRI as part of a neuroimaging sub-study (IRB# AAAO9758). Some participants (n=30) will already have had baseline amyloid PET imaging under PI IRB protocol # 7130R (BAY 949172PET/CT in Older Adults).
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
PET amyloid Standard Uptake Value ratio (SUVr) values | up to 18 months
  The primary outcome is the mean standard uptake value ratio in the 4 regions of interest.
Transcranial Doppler (TCD) dynamic autoregulatory dysfunction | up to 18 months
  Cerebral blood flow velocities (CBFV) are assessed using TCD. Arterial blood pressure (ABP) is recorded simultaneously using the Finapres on the middle phalanx of the left or right middle finger. The phase shift between the two streaming signals is an indication of the extent to which oscillations in CBFV lead those in ABP and can be interpreted as active early counter-regulation. Lower phase shift reflects increased latency in cerebral vasomotion and thus poorer autoregulation.

CONTACTS AND LOCATIONS:
Overall Officials: Adam M Brickman, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No